CLINICAL TRIAL: NCT03654833
Title: Mesothelioma Stratified Therapy (MiST): A Stratified Multi-arm Phase IIa Clinical Trial to Enable Accelerated Evaluation of Targeted Therapies for Relapsed Malignant Mesothelioma
Brief Title: Mesothelioma Stratified Therapy (MiST) : A Multi-drug Phase II Trial in Malignant Mesothelioma
Acronym: MiST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Collaborators: British Lung Foundation (Other); Clovis Oncology, Inc. (Industry); Eli Lilly and Company (Industry); Merck Sharp & Dohme LLC (Industry); BerGenBio ASA (Industry); Roche Pharma AG (Industry); University Hospitals, Leicester (Other); The Christie NHS Foundation Trust (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0627
Record Dates: First submitted 2018-08-07; First posted 2018-08-31 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-01

CONDITIONS: Mesothelioma, Malignant
Keywords: Drug: multi-arm; Phase IIa
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — rucaparib; abemaciclib; pembrolizumab; bemcentinib; atezolizumab; Bevacizumab; dostarlimab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MiST1 Rucaparib (Experimental): BRCA1/BAP1 negative mesothelioma; 600mg twice daily (BID) every 28 days.
  Interventions: Drug: Rucaparib
- MiST2 Abemaciclib (Experimental): p16INK4A negative mesothelioma; 200mg orally twice daily every 28 days.
  Interventions: Drug: Abemaciclib
- MiST3 Pembrolizumab & Bemcentinib (Experimental): No specific biomarker requirement: Pembrolizumab 200mg IV infusion on Day 1 only:
  Bemcentinib loading dose of 400mg on days 1-3, on day 4 on-wards 200mg daily every 21-days.
  Interventions: Drug: pembrolizumab & bemcentinib
- MiST4 Atezolizumab & Bevacizumab (Experimental): PDL1 expression positive mesothelioma: Atezolizumab 1200 milligrams via intravenous nfusion; Bevacizumab 15 milligrams per kilogram via IV infusion both on Days 1 every 21-days.
  Interventions: Drug: Atezolizumab & Bevacizumab
- MiST 5 Dostarlimab and Niraparib (Experimental): Platinum sensitive mesothelioma: Niraparib 200-300mg daily every 21 days; Dostarlimab 500mg on day 1 of each 21 day cycle for 4 cycles, then 1000mg on day 1 of each 42 day cycle.
  Interventions: Drug: Dostarlimab and Niraparib

INTERVENTIONS:
Drug: Rucaparib — PARP inhibitor
  Other Names: CO-338
  Arms: MiST1 Rucaparib
Drug: Abemaciclib — CDK4/6 inhibitor
  Other Names: LY2835219
  Arms: MiST2 Abemaciclib
Drug: pembrolizumab & bemcentinib — PD1 checkpoint inhibitor, AXL inhibitor
  Other Names: Keytruda; BGB324
  Arms: MiST3 Pembrolizumab & Bemcentinib
Drug: Atezolizumab & Bevacizumab — PDL1 checkpoint inhibitor, VEGF inhibitor
  Other Names: MPDL3280A; Avastin
  Arms: MiST4 Atezolizumab & Bevacizumab
Drug: Dostarlimab and Niraparib — IG Antibody, PARP Inhibitor
  Other Names: Zejula
  Arms: MiST 5 Dostarlimab and Niraparib

SUMMARY:
MiST is a British Lung Foundation funded, University of Leicester Study, a multi-arm stratified therapy based clinical trial for patients with relapsed mesothelioma.

The goal of MiST is to enable acceleration of novel, effective personalised therapy as a basis for improving survival outcomes for patients with mesothelioma.

DETAILED DESCRIPTION:
Stage 1 - molecular pre-screening:

The MiST Master protocol describes the identification of patients, biomarker testing and analysis. Patients with relapsed mesothelioma will be offered to consent for molecular panel testing of their diagnostic tumour block for predictive biomarkers. The results of this assessment will be used to classify patients into one of several possible molecularly defined treatment arms. Patients will therefore be offered a specific study treatment determined by their molecular profile. Patients, who exhibit positive testing in more than one biomarker, will potentially be eligible to subsequently be treated on a different treatment protocol upon disease progression or treatment failure.

Stage 2 - Treatment:

The MiST treatment protocol will be specific to the treatment allocated to the patient - based on the results of their biomarker testing in stage 1.

Specific agent(s) will be detailed separately in each of the separate treatment protocols.

Stage 3 - Molecular Profiling :

In order to understand the genomic basis of drug response in the MiST trial, archival tumour tissue from all patients enrolled will be interrogated using molecular inversion probe- based microarray analysis of the somatic copy number aberrations. Optional re-biopsy of patients who progress on treatment, followed confirmed radiological response, will be offered, to investigate genomic interrogation of tumours at the time of acquired resistance. For arms 3, 4 and 5 immune checkpoint, transcriptomic and gut microbiome correlative studies are planned.

ELIGIBILITY:
INCLUSION CRITERIA FOR PRE-SCREENING

* Histologically confirmed MM with an available biopsy for research purposes
* Male or female patients aged ≥18 years.
* Expected survival of ≥12 weeks or greater
* ECOG PS 0-1
* CT scan chest, abdomen (and pelvis if applicable) confirming disease progression.
* Patients must have received at least one prior line of therapy to include a platinum doublet first-line chemotherapy (within or outside of another clinical trial)
* Willing to consent for molecular screening of archived tumour block (PIS1 & CF1)

EXCLUSION CRITERIA FOR PRE-SCREENING

* Patients with a diagnosis of a second malignancy except prostate or cervical cancer in remission, patients with a diagnosis of basal cell carcinoma of the skin or superficial bladder cancer.
* Uncontrolled CNS disease. Asymptomatic brain metastases are allowed if previously treated with radiotherapy >28 days prior to starting the investigational agent.
* New York Heart Association Class II or greater congestive heart failure.
* Patients with severe hepatic insufficiency or severe renal impairment.
* Patients requiring long term oxygen therapy.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Each individual MiST drug protocol contains the eligibility criteria specific to the treatment allocated to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) at 12 weeks assessed by modified RECIST 1.1, in patients with relapsed mesothelioma. | 12 weeks
  This will be assessed using CT scan evidence according to modified RECIST 1.1 criteria reporting. Scans will be undertaken every 6 weeks. Analysis will be timed from study entry using the baseline CT scan results until completion of treatment cycles, confirmed disease progression or death - whichever comes first.

SECONDARY OUTCOMES:
Disease control rate (DCR) at 24 weeks assessed by modified RECIST 1.1, in patients with relapsed mesothelioma. | 24 weeks
  This will be assessed using CT scan evidence according to modified RECIST 1.1 criteria reporting. Scans will be undertaken every 6 weeks. Analysis will be timed from study entry using the baseline CT scan results until completion of treatment cycles, confirmed disease progression or death - whichever comes first.
Objective response rate (ORR) assessed for 12 months | Up to 12 months (up to 6 months during treatment and 6 months of follow-up)
  This will be assessed using CT scan evidence according to modified RECIST 1.1 criteria
Safety assessed according to CTCAE criteria. | 12 months (up to 6 months during treatment and 6 months of follow-up)
  Adverse events will be recorded in relation to each cycle of treatment and graded according to Common Terminology Criteria for Adverse Events (CTCAE). The incidence of each adverse event (all grades and grade 3/4) will be reported as a per-patient-cycle rate and as a per-patient rate. Investigators expect patients to participate in the study for a maximum of 6 months of Treatment and 6 months of follow-up, however cannot guarantee that some patients may participate over 12 months.
Toxicity assessed according to CTCAE criteria. | 12 months (up to 6 months during treatment and 6 months of follow-up)
  Adverse events will be recorded in relation to each cycle of treatment and graded according to Common Terminology Criteria for Adverse Events (CTCAE). The incidence of each adverse event (all grades and grade 3/4) will be reported as a per-patient-cycle rate and as a per-patient rate. Investigators expect patients to participate in the study for a maximum of 6 months of Treatment and 6 months of follow-up, however cannot guarantee that some patients may participate over 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fennell, PhD, FRCP, Study Director — University of Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fennell DA, King A, Mohammed S, Greystoke A, Anthony S, Poile C, Nusrat N, Scotland M, Bhundia V, Branson A, Brookes C, Darlison L, Dawson AG, Gaba A, Hutka M, Morgan B, Bajaj A, Richards C, Wells-Jordan P, Thomas A; MiST2 study group. Abemaciclib in patients with p16ink4A-deficient mesothelioma (MiST2): a single-arm, open-label, phase 2 trial. Lancet Oncol. 2022 Mar;23(3):374-381. doi: 10.1016/S1470-2045(22)00062-6. Epub 2022 Feb 11. PMID 35157829
- [Derived] Fennell DA, King A, Mohammed S, Branson A, Brookes C, Darlison L, Dawson AG, Gaba A, Hutka M, Morgan B, Nicholson A, Richards C, Wells-Jordan P, Murphy GJ, Thomas A; MiST1 study group. Rucaparib in patients with BAP1-deficient or BRCA1-deficient mesothelioma (MiST1): an open-label, single-arm, phase 2a clinical trial. Lancet Respir Med. 2021 Jun;9(6):593-600. doi: 10.1016/S2213-2600(20)30390-8. Epub 2021 Jan 27. PMID 33515503